CLINICAL TRIAL: NCT05191680
Title: Targeted Drug Intervention in Men at Risk of Progression on Active Surveillance for Early Prostate Cancer: A Randomised Trial - Therapeutics in Active Prostate Cancer Surveillance (TAPS02).
Brief Title: TherApeutics in Early ProState Cancer (TAPS02)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); Janssen-Cilag Ltd. (Industry)
Responsible Party: Principal Investigator, Vincent Gnanapragasam, Professor of Urology and Honorary Consultant Urologist, Cambridge University Hospitals NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TAPS02; 2021-006106-75 (EudraCT Number)
Record Dates: First submitted 2021-12-16; First posted 2022-01-13 (Actual); Last update posted 2025-06-20 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: active surveillance; prostate cancer; therapeutics in prostate cancer; apalutamide; short term androgen deprivation therapy; androgen receptor inhibitor
MeSH Terms: conditions — Prostatic Neoplasms | interventions — apalutamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Apalutamide 6 months (Experimental): Participants will receive apalutamide 240 mg (4 x 60 mg tablets) orally once a day for up to 6 months.
  Interventions: Drug: Apalutamide Oral Tablet [Erleada]
- Apalutamide 3 months + Placebo 3 months (Experimental): Participants will receive apalutamide 240mg (4 x 60 mg tablets) orally once a day for up to 3 months followed by placebo to match apalutamide (4 tablets) orally once a day for up to 3 months.
  Interventions: Drug: Apalutamide Oral Tablet [Erleada]; Drug: Placebo
- Placebo 6 months (Placebo Comparator): Participants will receive placebo to match apalutamide (4 tablets) orally once a day for up to 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Apalutamide Oral Tablet [Erleada] — Apalutamide is a selective Androgen Receptor (AR) inhibitor that binds directly to the ligand-binding domain of the AR.
  Other Names: Erleada
  Arms: Apalutamide 3 months + Placebo 3 months; Apalutamide 6 months
Drug: Placebo — Placebo to match apalutamide
  Arms: Apalutamide 3 months + Placebo 3 months; Placebo 6 months

SUMMARY:
This is a phase 2, randomised, multicentre, double-blind, placebo-controlled trial investigating the use of short term androgen deprivation therapy in the form of apalutamide (Erleada) in men on active surveillance for prostate cancer.

ELIGIBILITY:
INCLUSION CRITERIA

To be included in the trial the patient must:

* Have given written informed consent to participate.
* Be aged 18 or over.
* Have an Eastern Cooperative Oncology Group (ECOG) status 0-2.
* Have selected active surveillance as a management option.
* Have an MRI detectable lesion with an M score of ≥ 3 using Likert scale OR PI-RADS (version 2.1) reporting criteria. If M score is 3 then lesion size (single or combined) of ≥10mm.
* Have prostate cancer from a combination of image guided targeted + systematic biopsies and MRI lesion and biopsy are concordant for a prostate cancer diagnosis.
* Not anticipated to require bladder outlet surgery during IMP treatment or for up to 12 months of follow-up.
* Meet all of the following clinical laboratory assessment criteria:

  * Haemoglobin ≥ 9.0 g/dL, independent of transfusion and/or growth factors within 3 months prior to randomisation.
  * Platelet count ≥ 100 x 109/L independent of transfusion and/or growth factors within 3 months prior to randomisation.
  * Absolute neutrophil count (ANC) ≥ 1.0 x 109/L within 21 days prior to randomisation.
  * Serum albumin ≥ 3.0 g/dL within 21 days prior to randomisation.
  * Glomerular filtration rate (GFR) ≥ 30 ml/min AND Serum creatinine ≤ 3 times the ULN (calculated by Cockcroft and Gault equation using actual body weight) within 21 days prior to randomisation.
  * Serum potassium ≥3.5 mmol/L within 21 days prior to randomisation.
  * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤2.5 × ULN AND Serum total bilirubin ≤1.5 × ULN within 21 days prior to randomisation (Note: In patients with confirmed Gilbert's syndrome, if total bilirubin is >1.5 × ULN, measure direct and indirect bilirubin and if direct bilirubin is ≤1.5 × ULN, patient may be eligible in consultation with their physician).
* Have prostate cancer with any one or more of the following:

  * CPG2 (based on Grade Group 2 on histology)
  * CPG1 (based on Grade Group 1 on histology) with PSA high density (PSAd >0.15) and LIKERT or PI-RADS 4/5 lesion (individual or combined) of ≥10mm size.
  * CPG1 with PSA high density (PSAd >0.15) and ≥50% biopsy core involvement (number of positive cores/all cores taken) with target biopsies counted as one if LIKERT or PI-RADS 3 lesion

EXCLUSION CRITERIA

The presence of any of the following will preclude patient inclusion:

* Contraindications to apalutamide or its excipients.
* Pelvic metalwork interfering with MRI prostate interpretation.
* Any prior or concurrent use of androgen deprivation therapy (ADT) or androgen receptor targeting agents (not including established and continued use of 5-ARIs for urinary symptoms).
* Systemic therapy for prostate cancer.
* Inability for patient to have prostate MRI scan.
* Concurrent involvement in a Clinical Trial of Investigational Medicinal Product (CTIMP); participation in an observational trial/studies is acceptable.
* Seizure or known condition that may pre-dispose to seizure (including but not limited to the following within 1 year prior to randomisation: prior stroke, transient ischemic attack, loss of consciousness, brain arteriovenous malformation; or intracranial masses such as schwannomas and meningiomas that are causing oedema or mass effect).
* Medications known to lower the seizure threshold or cause seizures must be discontinued or substituted at least 28 days prior to randomisation.
* In the opinion of investigator, patient is at increased risk of falls or fractures.
* Severe/unstable angina, myocardial infarction, symptomatic congestive heart failure, arterial or venous thromboembolic events (e.g., pulmonary embolism, cerebrovascular accident including transient ischemic attacks), or clinically significant ventricular arrhythmias within 6 months prior to randomisation. Cardiovascular risk factors should be optimised i.e. hypertension, diabetes, dyslipidaemia.
* Uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 90 mmHg). Patients with a history of uncontrolled hypertension are allowed provided blood pressure is controlled by anti-hypertensive treatment.
* Gastrointestinal disorder affecting absorption.
* Medicinal products known to prolong the QT interval or medicinal products able to induce Torsade de pointes such as class IA (e.g., quinidine, disopyramide) or class III (e.g., amiodarone, sotalol, dofetilide, ibutilide) antiarrhythmic medicinal products, methadone, moxifloxacin, antipsychotics (e.g. haloperidol). Alternative therapy, for the prohibited medication known to prolong the QTc, may be inistigated. A minimum washout for the discontinued medication of ≥ 4 half-lives is required prior to starting IMP.
* Symptoms suggestive of Stevens-Johnson syndrome (SJS)/toxic epidermal necrolysis (TEN).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
MRI defined tumour volume | 12 months after end of treatment
  To determine whether there is a reduction in MRI defined tumour volume at 12 months post treatment in at least 50% of the treated cohort in either treatment arm compared to the baseline measurement.

SECONDARY OUTCOMES:
Reported adverse events | Reported from the point of obtaining informed consent until the safety FU visit (30-45 days post-treatment)
  As per NCI-CTCAE v5.0
Patient-reported outcomes EORTC QLQ-C30 | Cumulative until 12 months after end of treatment
  Assessed using the European Organisation for Research and Treatment of Cancer Quality of Life of Cancer Patients questionnaire (EORTC QLQ-C30).
Patient-reported outcomes EQ-5D-5L | Cumulative until 12 months after end of treatment
  Assessed using the EQ-5D-5L questionnaire developed by the EuroQol Group.
Cumulative rate of progression (any progression) | 3 years after completion of treatment
  the overall rate of disease progression
Cumulative rate of progression to any prostate cancer treatment (for any cause) | 3 years after completion of treatment
  the overall rate of conversion to treatment for any causes

CONTACTS AND LOCATIONS:
Overall Officials: Vincent J Gnanapragasam, Prof., Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (6):
- United Kingdom (6):
  - Addenbrooke's Hospital, Cambridge, Cambridgeshire
  - Southmead Hospital, Bristol
  - West Suffolk Hospital, Bury St Edmunds
  - Darent Valley Hospital, Dartford
  - St Bartholomew's Hospital, London
  - The Royal Marsden Hospital - Chelsea, London

IPD SHARING:
Plan to Share IPD: No